CLINICAL TRIAL: NCT05213455
Title: Booster Effect of mRNA Vaccine After Complete Vaccination With Sinos: an Observational Study
Brief Title: Booster Effect of mRNA Vaccine on Antibody Response for SARS-CoV-2 After Complete Vaccination With Sinos
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: LGH010
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: booster vaccine for COVID 19 — The effect of Booster vaccine will be seen in participants in terms of antibody response IgG

SUMMARY:
In most parts of the world, mRNA vaccines were used to provide protection to population against COVID 19. However, in some countries, including Pakistan, traditional viral vaccines named as Sinovac and Sinopharm were used for mass level immunization. Though these vaccines were approved by WHO, their efficacy had been questioned.

Now after recommendation of booster doses, we aim to see the effect of mRNA vaccine as a booster dose after Sinovac and Sinopharm in terms of antibody response. (IgG RBD SARS CoV2)

DETAILED DESCRIPTION:
In most parts of the world, mRNA vaccines were used to provide protection to population against COVID 19. However, in some countries, including Pakistan, traditional viral vaccines named as Sinovac and Sinopharm were used for mass level immunization. Though these vaccines were approved by WHO, their efficacy had been questioned.

Now after recommendation of booster doses, we aim to see the effect of mRNA vaccine (BNT162b2, pfizer) as a booster dose after Sinovac and Sinopharm in terms of antibody response. (IgG RBD SARS CoV2).

The antobody IgG RBD levels will be checked before the booster dose and then after 3 weeks of the booster.

ELIGIBILITY:
Inclusion Criteria:

* people who have received two doses of sinopharm or sinovac and six months have passed after the second dose

Exclusion Criteria:

* people getting one shot of sinopharm or sinovac or got vaccine other than sinopharm and sinovac.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include participants who have received two doses of sinopharm or sinovac and six months have passed after the second dose.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
IgG RBD levels | after 3 weeks of booster vaccine dose
  to see the effect of booster vaccine after 3 weeks in terms of IgG RBD

CONTACTS AND LOCATIONS:
Overall Officials: Amina Asif, M.Phil, Principal Investigator — Lahore General Hospital; Muhammad Irfan Malik, FRCP, Principal Investigator — Lahore General Hospital
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
will be available on request